CLINICAL TRIAL: NCT03439358
Title: Intravenous Magnesium Sulfate for the Prevention of Intraoperative Shivering in Parturients Undergoing Cesarean Delivery Under Lidocaine Top-up Via a Pre-existing Epidural Catheter Inserted for Labor Analgesia - A Randomized Double-blind, Placebo-controlled Trial
Brief Title: Magnesium for Shivering in Epidural Lidocaine Deliveries
Acronym: Mag-SHIELD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit patients
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H17-02408
Record Dates: First submitted 2018-02-07; First posted 2018-02-20 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia
Keywords: Epidural top-up; Shivering; Magnesium
MeSH Terms: interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulfate (Experimental): Magnesium sulfate (MgSO4) infusion will be commenced prior to epidural top-up.
  Interventions: Drug: Magnesium Sulfate
- Normal saline (Placebo Comparator): Normal saline infusion will be commenced prior to epidural top-up.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Magnesium Sulfate — Bolus infusion: 100mL normal saline with 4g MgSO4 over 30 minutes Maintenance infusion: 25mL normal saline per hour with 1g MgSO4
  Arms: Magnesium sulfate
Other: Normal Saline — Bolus infusion: 100mL normal saline over 30 minutes Maintenance infusion: 25mL normal saline per hour
  Arms: Normal saline

SUMMARY:
Magnesium has been shown to decrease the shivering experienced from neuraxial anesthesia. This study aims to investigate whether magnesium decreases the shivering experienced in parturients undergoing labor epidural anesthesia for Cesarean delivery.

DETAILED DESCRIPTION:
Women who have epidurals in place and go on to require a Cesarean delivery typically have their epidurals 'topped-up' with a fast onset local anesthetic to ensure the lower body is fully numb for surgery. This is called an epidural 'top-up'. However, a side effect of epidural top-ups is shivering, which is uncomfortable for the mother and interferes with patient monitoring. Magnesium administration has been shown to decrease shivering in the non-pregnant population. Therefore, in this study the investigators aim to determine if magnesium given prior to an epidural top-up decreases the incidence and severity of shivering in the pregnant population.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age of ≥37 weeks
2. Women who are ≥ 19 years old
3. Women undergoing Cesarean delivery under lidocaine top-up via a preexisting epidural catheter inserted for labor analgesia
4. American Society of Anesthesiologist (ASA) Physical Status class 1 or 2

Exclusion Criteria:

1. Emergency Cesarean delivery with limited time for informed consent
2. Women who have received MgSO4 prior to study enrollment
3. Indication for alternative mode of anesthesia for Cesarean delivery (e.g., general anesthesia)
4. Medical conditions or medications that could lead to tremor or shivering. (e.g., movement disorder, untreated thyroid disease) or mask tremor or shivering (e.g., beta-blocker, benzodiazepine, anticonvulsants)
5. Active shivering at time of recruitment
6. Inability to read and understand English for the purpose of informed consent
7. Contraindications to receiving MgSO4 (hypersensitivity reactions, respiratory rate <16breaths/min, absent reflexes, urine output <100 mL during the previous 4 hours, renal failure, or hypocalcemia)
8. History of previous postpartum hemorrhage

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative shivering | Through completion of cesarean surgical procedure (maximum 2 hours)
  Incidence measured as shivering present or absent
Severity of intraoperative shivering | Through completion of cesarean surgical procedure (maximum 2 hours)
  Severity measured subjectively by anesthesiologist and patient

SECONDARY OUTCOMES:
Incidence of hypothermia | Through study completion (maximum 2.5 hours)
  Number of patients whose tympanic membrane temperature decreases below 36 degrees Celsius.
Incidence of hypotension | Through study completion (maximum 2.5 hours)
  Number of patients who experience a greater than or equal to 20% reduction in systolic blood pressure.
Total vasopressor(s) dose | Through study completion (maximum 2.5 hours)
Total utertonic(s) dose | Through completion of cesarean surgical procedure (maximum 2 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD MMSc, Principal Investigator — University of British Columbia; Anna West, BA MBBS, Study Chair — University of British Columbia; Vit Gunka, MD, Study Chair — University of British Columbia; Jonathan Collins, BA BM BCh MA, Study Chair — University of British Columbia; Monica Brunner, MD, Study Chair — University of British Columbia; Arianne Albert, PhD, Study Chair — Provincial Health Services Authority British Columbia; James D Taylor, BSc, Study Chair — Provincial Health Services Authority British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No